CLINICAL TRIAL: NCT03320889
Title: Hepatitis C Education for Pregnant Women With Opiate Dependence - Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-057
Record Dates: First submitted 2017-10-02; First posted 2017-10-25 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Group 1: Educational Intervention includes Pamphlets plus Review with Expert Educator Group 2: Educational Intervention includes Pamphlets only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pamphlets plus Review with Expert Educator (Other): Educational Intervention includes Pamphlets plus Review with Expert Educator
  Interventions: Other: Educational Intervention
- Pamphlets only (Other): Educational Intervention includes Pamphlets only
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Patients will be randomized to a group that receives the pamphlets only and a group that receives the pamphlets and has an expert educator review that pamphlets with them and answer questions.

SUMMARY:
The goal of this study is to assess patients' attitudes and knowledge of Hepatitis C, analyze the variables that may influence patients' knowledge, and educate patients on Hepatitis C.

DETAILED DESCRIPTION:
The study will compare the effectiveness of providing HCV education by providing a pamphlet and expert education compared to providing a pamphlet only. The information gained in completing this study will help the medical community improve patient education on the disease and specifically understand how the medical community can best serve pregnant patients with opiate dependence burdened by Hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Study population includes Faculty Medical Center obstetrics and postpartum patients enrolled in the HOPE program who are 18 years old or older.
* The study will include patients with and without a Hepatitis C diagnosis.
* Patients will be recruited at their routine office visits and/or during any admissions to the hospital.

Exclusion Criteria:

* Patients who do not speak and understand English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Number of Questions Scored Correct on the Hepatitis C Knowledge Survey | 2-8 weeks after study intervention
  Number of questions scored correct on the Hepatitis C knowledge survey

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marcotte, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No